CLINICAL TRIAL: NCT02905994
Title: A Phase I Trial of Volasertib (BI 6727), an Intravenous Polo-Like Kinase Inhibitor, in Combination With "7+3" Induction Chemotherapy for Patients With Acute Myeloid Leukemia
Brief Title: Volasertib Combined With Induction Chemotherapy in Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding Withdrawn
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Amir Fathi, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-299
Record Dates: First submitted 2016-09-12; First posted 2016-09-19 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: AML
Keywords: Leukemia
MeSH Terms: conditions — Leukemia | interventions — BI 6727; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volasertib with chemotherapy (Experimental): Patients enrolled on this trial will receive induction chemotherapy with "7+3"
  * Cytarabine continuous infusion days 1-7
  * Idarubicin IV bolus on days 1, 2, and 3.
  * Patients will receive Volasertib as an intravenous infusion over approximately 1 hour, according to dosing level, on day 8
  * Patients will receive Standard Anti Fungal and Standard Antibiotic during induction
  * A bone marrow biopsy will be performed according to standard practice on day 14
  Interventions: Drug: Volasertib; Drug: Cytarabine; Drug: Idarubicin; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Drug: Volasertib — Polo-Like Kinase Inhibitor
  Other Names: BI 6727
Drug: Cytarabine — Standard chemotherapy at dosage and schedule for 7+3 induction
  Other Names: Depocyt
Drug: Idarubicin — Standard chemotherapy at dosage and schedule for 7+3 induction
  Other Names: Idamycin
Procedure: Bone Marrow Biopsy — Bone marrow biopsy assessments scheduled during induction to assess response

SUMMARY:
The study intervention involved in this study is the addition of a dose of volasertib as a part of the initial chemotherapy regimen for AML.

The trial will involve a combination of the following drugs:

* Volasertib (the study drug)
* Idarubicin
* Cytarabine

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

As part of this research study, the participant will receive Volasertib in combination with two other chemotherapy drugs, Idarubicin and Cytarabine. The FDA (the U.S. Food and Drug Administration) has not approved volasertib as a treatment for any disease.

Idarubicin and Cytarabine are chemotherapy agents that are commonly used to treat individuals diagnosed with AML. Volasertib inhibits proteins called "polo-like kinases," which are necessary for cell division. Volasertib binds to these proteins and this inhibits the growth of cancer cells. Volasertib has been used in laboratory studies and those studies suggest that volasertib may slow down the growth of Cancer. In a previous clinical trial in patients with the participant type of leukemia where Volasertib was given along with low doses of Cytarabine, this drug was found to have some clinical activity against AML. In this study, researchers would like to combine Volasertib with standard chemotherapy (Cytarabine and Idarubicin) in order to see if it can be given safely with chemotherapy in individuals with AML.

The primary purpose of this research study is to determine the highest dose that Volasertib can be given with Idarubicin and Cytarabine without severe or unmanageable side effects. The dose identified in this study will be used in future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed, newly diagnosed acute myeloid leukemia.
* Adults, age 18 years or older at the time of diagnosis, eligible for standard induction chemotherapy according to their treating physician.
* ECOG performance status 0-2 (Karnofsky ≥60%, see Appendix A)
* Left ventricular ejection fraction > 50% as measured by echocardiogram or MUGA scan
* Must not have received systemic antineoplastic therapy including radiation therapy within 14 days of the study enrollment, except hydroxyurea or 6-mercaptopurine for the purposes of cytoreduction as per the treating physician. Patients may also have received all-trans retinoic acid (ATRA) if there is an early suspicion of acute promyelocytic leukemia (APL, M3-AML), although if confirmed to have APL these patients will be excluded from the study.
* Female patients of childbearing age must have negative pregnancy test.
* Participants must have normal organ and marrow function as defined below:

  * total bilirubin < 3 times the ULN
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of volasertib (BI 6727) on the developing human fetus are unknown. For this reason and because other chemotherapeutic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and 6 months after completion of therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and 6 months after completion of therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients will be excluded from this study if they are found to harbor "favorable" risk cytogenetics41 including:

  * APL, t(15;17)
  * t(8;21)
  * inv(16) or t(16;16) A sample to evaluate patient cytogenetics will be sent at the time of diagnosis per standard clinical care and the absence of these cytogenetics must be confirmed by Day 8. If the cytogenetic analysis reveals that the patient harbors favorable risk cytogenetics, or if the cytogenetic results are not received prior to Day 8, the participant will be removed from the study.
* Patients with acute bilineal/biphenotypic leukemia
* Participants who have had chemotherapy or radiotherapy within 14 days prior to entering the study, except for hydroxyurea, 6-MP, and ATRA, as noted.
* Participants who are receiving any other investigational agents.
* Chemo-, hormono-, radio- or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug
* Persistence of clinically relevant therapy related toxicity from previous anti-cancer therapy
* Prior allogeneic bone marrow or organ transplantation
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Current clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukemic CNS involvement (no lumbar puncture required, clinical assessment per investigator's judgment is sufficient).
* Prior treatment with volasertib or another polo-like kinase inhibitor
* A diagnosis of active Hepatitis B or C infection. A patient with a prior infection may participate, so long as the infection is not active at the time of study screening tests and according to investigator discretion.
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome. Baseline QTc must be 470 msec or less, according to the Friderica correction method,42 calculated as the mean of 3 ECGs taken at the time of screening.
* Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF <50%, as measured by MUGA scan or echocardiogram).
* Known hypersensitivity to the trial drugs or other contraindication to standard "7+3" induction chemotherapy.
* Although not absolute exclusion criteria, several known drug-drug interactions should be considered during enrollment (see Section 5.5).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because volasertib, along with standard induction chemotherapy, carries the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with volasertib as well as cytarabine and idarubicin, breastfeeding should be avoided.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with volasertib. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
* Patients who are otherwise felt unable to comply with the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Establishing The Maximum Tolerated Dose (MTD) | 2 years

SECONDARY OUTCOMES:
Rate of Complete Response | 2 years
Rate of Relapse Free Survival | 1 year
Rate of Overall Survival | 1 year
Rate of partial response | 2 years
Degree of change in the presence of subclones with Disease Response | 2 years
  Measured by subclonal disease evolution, during treatment with volasertib and "7+3"
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amir T Fathi, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts general Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No